CLINICAL TRIAL: NCT07382310
Title: Effect of Different Products to Support Plaque Control During Daytime: a Cross-over Single Blinded Randomized Controlled Clinical Trial
Brief Title: Effect of Different Products to Support Plaque Control During Daytime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: The University of Sydney, Sydney, Australia (Unknown)
Responsible Party: Principal Investigator, Lana Bader, Assistant professor, King Abdullah University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: X20-0076; X20-0076 - 2020/STE00758 (Other: Sydney Local Health district, Research Goverance office. Site specific approval at The Sydney Dental Hospital); X20-0076 - 2020/ETH00407 (Other: Ethics Review Committee (Royal Prince Alfred Hospital RPAH Zone) of the Sydney Local Health District)
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Dental Plaque; Dental Plaque Accumulation; Mouthwashes; Chewing Gum
Keywords: Dental plaque; Listerine Go tablet; Listerine Total care mouth wash; Oral B Pro-Health Multi-Protection Mouth Rinse; Colgate total advanced pro-shield mouth rinse; Wrigley Extra chewing gum; xylitol chewing gum
MeSH Terms: conditions — Dental Plaque | interventions — Ethanol; cytidylyl-(3'-5')-cytidine

STUDY DESIGN:
Intervention Model Description: Crossover, single blinded, randomised controlled clinical trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: All the assessed parameters were measured by one examiner (L.B) who was blinded. A hospital staff member (dental hygienist, F.Z) was responsible for giving the products to the participants. Each participant was given a unique serial identification number composed of two digits. A unique study ID was used to link participants' name, photos, and product used. The hygienist kept a sheet for each participant. On that sheet the following information was recorded:
  * Unique study ID for each participant.
  * Participant's first name, surname and date of birth.
  * Computer generated randomisation list of control and tested products marked as: product A, product B ... etc.
  * The date when each product was disposed to the participant and the type of product.
  On each experiment day, a sticker was generated to include the unique ID and the product code that supposed to be received on that day (such as: PPCS 1 Product A, PPCS 2 Product B…etc). It was used to link the oral photos to the unique ID.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Listerine Total Care mouth rinse without alcohol (Active Comparator): Participants need to use the mouth wash twice a day (after tea break and after lunch break) according to manifacturer instructions: vigorously swish 20mL of rinse in your mouth for 30 seconds and then spit out. Do not swallow. Do not dilute. They were dispensed in their original bottles. Participants were given a marked cup to measure the amount of MW.
  Interventions: Drug: Listerine Total Care mouth rinse without alcohol
- Oral B Pro-Health Multi-Protection Mouth Rinse refreshing mint without alcohol (0.07% CPC) (Active Comparator): Participants need to use the mouth wash twice a day (after tea break and after lunch break) according to manifacturer instructions: vigorously swish 20mL of rinse in your mouth for 30 seconds and then spit out. Do not swallow. Do not dilute. They were dispensed in their original bottles. Participants were given a marked cup to measure the amount of MW.
  Interventions: Drug: Oral B Pro-Health Multi-Protection Mouth Rinse refreshing mint without alcohol (0.07% CPC)
- Colgate total advanced pro-shield mouth rinse without alcohol (0.075% CPC) (Active Comparator): Participants need to use the mouth wash twice a day (after tea break and after lunch break) according to manifacturer instructions: vigorously swish 20mL of rinse in your mouth for 30 seconds and then spit out. Do not swallow. Do not dilute. They were dispensed in their original bottles. Participants were given a marked cup to measure the amount of MW.
  Interventions: Drug: Colgate total advanced pro-shield mouth rinse without alcohol (0.075% CPC)
- Listerine Go Tabs (Active Comparator): Participants need to use the tablet twice a day (after tea break and after lunch break) according to manifacturer instructions: chew for 10 seconds to activate, swish around the teeth for 30 seconds to clean then swallow.
  Interventions: Drug: Listerine Go Tabs
- Wrigley Extra White Soft Chew Peppermint chewing gum. (Active Comparator): Participants need to use the chewing gum twice a day (after tea break and after lunch break) for 10 minutes duration.
  Interventions: Drug: Wrigley Extra White Soft Chew Peppermint chewing gum.
- Control (No Intervention): Participants will not recieve any product to use on the control day

INTERVENTIONS:
Drug: Oral B Pro-Health Multi-Protection Mouth Rinse refreshing mint without alcohol (0.07% CPC) — Participants need to use the mouth wash twice a day (after tea break and after lunch break) according to manifacturer instructions: vigorously swish 20mL of rinse in your mouth for 30 seconds and then spit out. Do not swallow. Do not dilute. They were dispensed in their original bottles. Participants were given a marked cup to measure the amount of MW.
  Arms: Oral B Pro-Health Multi-Protection Mouth Rinse refreshing mint without alcohol (0.07% CPC)
Drug: Listerine Total Care mouth rinse without alcohol — Participants need to use the mouth wash twice a day (after tea break and after lunch break) according to manifacturer instructions: vigorously swish 20mL of rinse in your mouth for 30 seconds and then spit out. Do not swallow. Do not dilute. They were dispensed in their original bottles. Participants were given a marked cup to measure the amount of MW.
  Arms: Listerine Total Care mouth rinse without alcohol
Drug: Colgate total advanced pro-shield mouth rinse without alcohol (0.075% CPC) — Participants need to use the mouth wash twice a day (after tea break and after lunch break) according to manifacturer instructions: vigorously swish 20mL of rinse in your mouth for 30 seconds and then spit out. Do not swallow. Do not dilute. They were dispensed in their original bottles. Participants were given a marked cup to measure the amount of MW.
  Arms: Colgate total advanced pro-shield mouth rinse without alcohol (0.075% CPC)
Drug: Listerine Go Tabs — Participants need to use the tablet twice a day (after tea break and after lunch break) according to manifacturer instructions: chew for 10 seconds to activate, swish around the teeth for 30 seconds to clean then swallow.
  Arms: Listerine Go Tabs
Drug: Wrigley Extra White Soft Chew Peppermint chewing gum. — Participants need to use the chewing gum twice a day (after tea break and after lunch break) for 10 minutes duration.
  Arms: Wrigley Extra White Soft Chew Peppermint chewing gum.

SUMMARY:
The goal of this clinical trial is to test if the additional use of different commercially available products for a better breath and plaque reduction, taken during daytime between morning and evening tooth brushing, can reduce the plaque formation of participants during the day.

The tested products were:

* Listerine Total Care mouth rinse without alcohol.
* Oral B Pro-Health Multi-Protection Mouth Rinse refreshing mint without alcohol.
* Colgate total advanced pro-shield mouth rinse without alcohol.
* Listerine Go Tabs.
* Wrigley Extra White Soft Chew Peppermint chewing gum.

The main questions it aims to answer are:

Can the tested product lower the plaque formation? Can the tested product improve the mouth freshness and breath?

Researchers will compare the tested products to not using any product (controls).

Participants need to come for a screening appointment and sign a consent form at first. If they are eligible, they need to come 6 times to the clinic. On each day, they need to come twice (morning appointment at 8 a.m. and evening appointment at 4 p.m.).

In the morning, they will have teeth cleaning and recieve one of the tested products to use on that day only (after tea break and lunch break), or they will recieve no product (control day).

In the evening, participant's teeth will be stained and oral photos will be taken. They will be asked about their perciption of freshness and good breath after using the product.

DETAILED DESCRIPTION:
Sample size, study location, and target population:

By using t-test and assuming a pooled standard deviation of 0.35 units, the study required a sample size of 15 participants in total, to achieve a 90% power and 1% level of significance (P<0.05), for detecting a true difference in means between the test and the control group of 0.5 on RMNPI index (Cugini et al 2006). This study is a cross-over study. In other words, participants were their own controls. Therefore, a total number of twenty participants were included in the study (10 males and 10 females).

The staff members of Sydney Dental Hospital were contacted by email to participate in the study. A screening appointment was arranged for interested participants to check for the eligibility criteria.

Study protocol:

One examiner (L.B) examined all participants two or three days a week. One participant was assessed per day. All eligible participants attended the Sydney Dental Hospital for 6 days. On each day, each participant was given a product to use on that day only according to the participant's own randomization list of products. If the day was a control day according to the participant's specific sheet, the participant did not receive anything. Then, the date was documented on each subject's own sheet. A minimum of 3 days wash out period was allowed between experimental days.

The following procedures were performed on each day:

On the control day (no products were used on that day): participants attended one morning appointment (at 8 a.m.) and one evening appointment (at 4 p.m.). Each appointment was about 45 min long.

* In the morning appointment: a disclosing agent (GC Tri Plaque Id Gel: GC America) was used to stain plaque. Then, all participants received a standardized full mouth professional prophylaxis and cleaning using Airflow Prophylaxis Master including Airflow hand piece with erythritol powder and Piezon handpiece to remove any hard deposits if needed (EMS, Switzerland). At that stage, clinical intra-oral photos were taken for all teeth surfaces using the Periodontic Department digital camera (Canon) to show that the mouth is 100% clean. As this is a control day, participants did not receive any of the tested products to be used on that day. They were allowed to practice their normal behaviour during daytime, but they were refrained from brushing, flossing or doing any oral hygiene practice until their evening appointment.
* In the evening appointment: the same disclosing agent was used to stain plaque and clinical intra-oral photos were taken for all teeth surfaces to measure RMNPI. This allowed plaque accumulation for about 7 hours. After that, all participants received the same full mouth professional prophylaxis and cleaning to obtain plaque free mouth.

On the other test days (participants received one test product on each day to use for that day only): similar to the control day, participants had to attend one morning appointment (at 8 a.m.) and one evening appointment (at 4 p.m.). Each appointment was about 45 min long.

* In the morning appointment: the same as the control day was done. In addition, each participant received one of the tested products on each day, according to a computer-generated randomization sequence, to test its effect for that day only. Each product was used twice a day: after tea break at 11 a.m. and after lunch break at 2 p.m., allowing 7 hours of plaque accumulation. Participants' compliance was self-reported. The Products were used according to manufacturer instructions as follows:

  * Mouth washes: Vigorously swish 20mL of rinse in your mouth for 30 seconds and then spit out. Do not swallow. Do not dilute. They were dispensed in their original bottles. Participants were given a marked cup to measure the amount of MW.
  * Listerine Go Tab: Chew for 10 seconds to activate, swish around the teeth for 30 seconds to clean then swallow.
  * Chewing gum: no manufacturer recommendation for the chewing duration, so as done in previous studies, 10 minutes duration was standardized for the chewing duration.
* In the evening appointment: same as control day was done. In addition, VAS was used to record participants' perception of fresh breath and cleanness in their mouth after using the product.

After all participants completed their visits, all photos were assessed to score RMNPI. All data were recorded on an excel sheet that was used to perform the statistical analysis.

Statistical analysis:

Statistical Analysis was conducted using SAS OnDemand for Academics (SAS Institute Inc., Cary, NC, USA). Data was checked for normality using Shapiro-Wilk test. As data proved non-homogeneous and not-normally distributed, Non-parametric Mann-Whitney U test was used to compare medians between groups (pair-wise), and Kruskal Wallis test for multiple groups comparisons. Pair-wise comparisons of significant differences in Kruskal Wallis test were made using the rank-transformed data using Tukey's adjustment to control for type I error. The results in tables are presented as Medians (95% confidence interval). Any differences were considered significant at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age is 18 years or more.
* Generally healthy.
* All teeth (28 teeth, excluding 3rd molars) should be present.
* The absence of untreated caries, secondary caries or faulty restorations.
* No orthodontic appliances (removable or/and fixed).
* No oral lesions, no active periodontal disease (no active inflammation or bleeding).
* Not using a mouthwash or any chewing product in the last week before the beginning of the study.

Exclusion Criteria:

* Pregnancy, lactation.
* Any chronic disease including diabetes, cardiac disease and diseases of the immune system.
* Presence of signs and symptoms of an acute infection in the oral cavity.
* Any prescribed systemic or topical medication.
* Any known allergies against ingredients of the different tested products.
* Use of antibiotics in the last 3 months.
* Use of nonsteroidal anti-inflammatory drugs (NSAID) in the last 3 months.
* History of alcohol or drug abuse.
* Smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Plaque index | At the end of each test day (6 days)
  Plaque accumulation assessed using the Rustogi Modified Navy Plaque Index (RMNPI) on designated tooth surfaces in the sides assigned to interdental brush and water flosser. The tooth was divided into multiple zones as the following :
  Whole mouth: areas A,B,C,D,E,F,G and H. Marginal (gum line): areas A,B and C. Interproximal: areas D and F
  0 score was given the area where there is no plaque.
  1 score was given in the area where there is plaque The minimum plaque score per surface (buccal or lingual) is zero, and the maximum plaque score per surface is 8 Intraoral photos using professional camera were taken for all teeth and all surfaces to record the plaque score.

SECONDARY OUTCOMES:
Patient reported outcome using visual analoge scale (VAS) | The VAS was reported by the patients at the end of the assessment day (6 days)
  The perception of cleanness, freshness, and good breath was measured on a visual analogue scale (VAS) from 0 - 10 (0 - being no clean feeling, no freshness or good breath. 10 - feeling of a very clean and fresh mouth with a good breath).

CONTACTS AND LOCATIONS:
Overall Officials: Axel Spahr, Study Director — University of Sydney; Lana Bader, DClinDent Perio, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Sydney Dental Hospital (SDH), Sydney, New South Wales, Central, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for plaque index (RMNPI) and patient-reported outcomes will be shared. Data will be stripped of all identifiers to protect participants privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD and supporting documents will be available after publication of the main study results, for a period of one year, starting from the day of research publication.
Access Criteria: Access will be granted to qualified researchers who request the data via email to the principal investigator. Researchers must sign a data use agreement ensuring ethical use, confidentiality, and prohibition of attempts to identify participants.